CLINICAL TRIAL: NCT02328651
Title: Effect and Safety of Xiao'er Jiebiao Oral Liquid in Combination With Standard Treatment on Hand-foot-mouth Disease in Pediatric Patients
Brief Title: Effect of Xiaoer Jiebiao Oral Liquid on Hand-foot-mouth Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Weihai Rensheng Pharmacy (Unknown)
Responsible Party: Principal Investigator, Hui Yu, Professor, Director, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XEJB_Ver1.0
Record Dates: First submitted 2014-12-18; First posted 2014-12-31 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Handfoot-mouth Disease
Keywords: Mild and Moderate Severe Patients With hand_foot-mouth Disease
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Ribavirin

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Ribavirin treatment plus testing drug (Experimental)
  Interventions: Drug: Ribavirin plus Xiao'er jiebiao oral liquid
- Ribavirin treatment (Active Comparator)
  Interventions: Drug: Ribavirin

INTERVENTIONS:
Drug: Ribavirin plus Xiao'er jiebiao oral liquid — For mild (Phase I) patients: recommended treatment according to naitonal guildeline for treatment of mouth-foot-hand diseases 2010, including ①treatment for control symptoms ② ribavirin 15mg/kg/d（ diluted in 100ml 5%GS），qd, ivgg, in combination using of Xiaoer jiebiao oral liquid 5 ml, bid for children aged 1-2 years, tid for children aged 3-5 years.
  For moderate (Phase II) patients:
  recommended treatment according to naitonal guildeline for treatment of mouth-foot-hand diseases 2010, including ①treatment for control symptoms ② ribavirin 15mg/kg/d（ diluted in 100ml 5%GS），qd, intravenous drip, in combination using of Xiaoer jiebiao oral liquid 5 ml, bid for children aged 1-2 years, tid for children aged 3-5 years.③anti-intracranial pressure treatment: mannitol 2~5ml/kg,iv, Bid~tid）
  Arms: Ribavirin treatment plus testing drug
Drug: Ribavirin — For mild (PhaseI) patients : recommended treatment according to naitonal guildeline for treatment of mouth-foot-hand diseases 2010, including ①treatment for control symptoms ② ribavirin 15mg/kg/d（ diluted in 100ml 5%GS），qd, intravenous drip.
  For moderate (PhaseII) patients: recommended treatment according to naitonal guildeline for treatment of mouth-foot-hand diseases 2010, including ①treatment for control symptoms ② ribavirin 15mg/kg/d（ diluted in 100ml 5%GS），qd, intravenous drip, in combination using of Xiaoer jiebiao oral liquid 5 ml, bid for children aged 1-2 years, tid for children aged 3-5 years.③anti-intracranial pressure treatment: mannitol 2~5ml/kg, iv, Bid~tid）
  Arms: Ribavirin treatment

SUMMARY:
This is a single-blinded randomized trial aiming to evaluate the effectiveness of Xiaoer Jiebiao Oral liquid in combination with Ribavirin treatment on patients with hand-foot-mouth disease compared with the controlgroup that recieve only libavirin treatment.

ELIGIBILITY:
Inclusion Criteria:subjects should meet all of the following

* diagnosed as hand-foot-mouth disease grade I or grade II;
* body temperature at admission T>38℃，fever length<48 hours;
* no need for hormonotherapy or immunoglobulin therapy.
* signed written informed consent form

Exclusion Criteria:subjects should be excluded if meet any of the following

* with history of any heart, lung, kidney or liver diseases; under any hormonotherapy, immunoglobulin therapy or any other therapy.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2018-04-30 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Time (hours) taken from treatment start till body temperature dropping to normal | time length( hours) from treatment starting to the time that body temperature drop to normal 37.0 degree for 12 hours
Time (hours) taken from disease onset till body temperature dropping to normal | time length (hours) from the disease onset (the starting of fever) till the time that body temperature dropped to normal (37.0 degree) and lasting for at least 12 hours
Top body temperature at the 24th hour, 48th hour and the 72th hour from treatment starting. | from starting of treatment to the 24th hour, 48th hour, and the 72th hour
  top body temperature at 3 time points after treatment diarrhea

SECONDARY OUTCOMES:
adverse digestive tract symptoms | from start of treatment to discharge
  proportion of patients with digestive tract symptoms during treatment, such as vomit, abdomial pain or diarrhea
abnormal blood routine | from the start of treatment to discharge test
  defined as 1 if any abnormal blood routine occur, otherwise defined as 0
abnormal Urine routine | from the start of treatment to discharge
  defined as 1 if any liver function examination or kidney function examination occur, otherwise defined as 0

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China